CLINICAL TRIAL: NCT05398354
Title: Active Retirement: Effects of the Application of a Training Program on the Stimulation of the Sensory Motor System
Brief Title: Active Retirement: Effects of the Application of a Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Carolina Alexandra Cabo, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21040
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Training; Sensorimotor Disorder
Keywords: aging; quality of life; sensory motor; training

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization is performed using a random selection method from the waiting list and the data will be coded and transferred to the database, depending on the intervention group and control group. Data analysis will be done statistically.
  Each participant will be randomly assigned to each group after signing the informed consent and conducting the initial assessments. All laboratory samples and data collected will be identified with identification ID, safeguarding the confidentiality of the collected data.
  At the end of this study, all participants of the control group will be offered the same intervention as the exercise group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Retirement - intervention (Experimental): The duration of the program is 24-weeks, 2-times a week, for up to 50 minutes per session. The sessions will be divided into three phases: the initial phase (10 minutes) will consist of a 5-minute walk followed by a joint warm-up; fundamental phase (25 minutes) will work in an exercise circuit, this circuit will consist of 4 cycles, with 8 exercises each, with a duration of 50 seconds and a rest of 15 seconds, for the exchange of exercise; and return to calm (10 minutes), where we will perform muscle stretching.
  Interventions: Behavioral: Active retirement
- Active Retirement - control (No Intervention): The control group will only carry out the assessments and will be offered the same intervention as the intervention group at the end of the intervention.

INTERVENTIONS:
Behavioral: Active retirement — During the intervention, the sensorimotor training program will have a progressive increase in load, the exercises will be divided into 3 levels of intensity: easy (without external load, during the first 8 weeks), intermediate (application of external load: elastic bands, shin guards and free weights, from the 9th to the 16th week) and advanced (increased external load compared to the previous level, from the 17th to the 24th week).
  During the sessions we will still assess the intensity through the subjective perception of effort (RPE) scale. In addition, adherence and control of the level of control through the Physical Activity Enjoyment (PACES) survey applied to participants.
  Arms: Active Retirement - intervention

SUMMARY:
The study will include 160 participants. They will be randomized into 2 groups, experimental and control. The intervention will take place over 24 weeks. Parameters of body composition, quality of life, physical activity, strength, flexibility, postural control, gait, agility and execution speed will be determined.

DETAILED DESCRIPTION:
The intervention study will have a quasi-experimental, longitudinal and controlled design. The sample will participate in a supervised training program lasting 24 weeks, followed by a 1-year follow-up period. The sample will be divided into two groups, intervention group and control group.

The variables under study are physical activity in the last week; quality of life; lower and upper limb strength; flexibility of the lower and upper limbs; postural control; march; agility and execution speed. These variables will be evaluated in 4 moments: before the beginning of the training program; after 24 weeks of the program; after 6 months from the end of the program; and after 1 year.

A convenience sample will be recruited in the community of Almada, in partnership with the Municipality of Almada (CMA). The sample will be recruited according to the following inclusion criteria: residents in the municipality of Almada, individuals between 55 and 80 years of age, healthy people, who do not have prostheses (with the exception of dental prostheses), who have not undergone operations for over 6 months, and who can walk independently for up to 10 minutes. Participants will not be eligible if they are younger than 55 years of age or older than 80 years of age, have a musculoskeletal or neurological diagnosis and report a clinical cardiovascular diagnosis. Gender is not an exclusion criterion.

The training program will be carried out over a period of 24 weeks, with exercise sessions twice a week, lasting approximately 45 minutes each. The sessions were divided into three phases: initial phase; fundamental phase; and return to calm. Throughout the intervention, the sensorimotor training program will have a progressive increase in load, the exercises will be divided into 3 levels of intensity: easy, intermediate and advanced.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 55 years and 80 years;
* Agree to participate in the study;
* Healthy people;
* People without prostheses (with the exception of dental prostheses);
* People who have not been operated on for less than 6 months.

Exclusion Criteria:

* People with musculoskeletal diagnosis;
* People with problems in locomotion;
* Psychiatric diseases and neurological disorders;
* People with a clinical cardiovascular diagnosis.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Body weight | 1 year
  Weight evaluation will be done using a scale
Height | 1 year
  Height evaluation will be done using a stadiometer
Lower limbs muscle strength | 1 year
  Lower limbs muscle strength will be evaluated with chair stand-up test
Upper limbs muscle strength | 1 year
  The muscle strength of the upper limbs will be evaluated by forearm flexion test
Lower limbs flexibility | 1 year
  Lower limbs flexibility will be evaluated through the "sit and reach"
Upper limbs flexibility | 1 year
  The flexibility of the upper limbs will be assessed through "reaching behind the back"
Postural control | 1 year
  Postural control will be assessed using a force platform (Bertec4060-Columbus; USA). The evaluation will consist of measuring the oscillations in a static bipedal position, with eyes open (2 minutes) and with eyes closed (2 minutes).
Gait | 1 year
  Gait will be evaluated using the mobile application "phyphox" on the inner edge of the tibia, on the surface of the skin, to quantify the number of steps and time), participants will be asked to walk a pre-established route, without slopes or obstacles, for 10 minutes at its natural cadence and then the same route at a rhythm determined by complex stimuli (auditory metronome - loudspeakers, which allow you to hear the beats, where each beat corresponds to a step)
Agility and execution speed | 1 year
  Agility and speed of execution will be evaluated through the application of the Timed Up and Go (TUG) test, which consists of getting up from a chair, walking to a straight line 3 meters away, turning, walking back and sitting down again.

SECONDARY OUTCOMES:
Life Quality | 1 year
  Quality of life will be assessed using the general health and well-being questionnaire. The questionnaire consists of 11 questions ranging from 1 to 5, where 1 is absolutely true and 5 is absolutely false.
Physical activity level | 1 year
  The practice of physical activity will be evaluated through the International Physical Activity Questionnaire. It does not have minimum and maximum values, the participants only indicate if they take place and in what period of time.
Effort intensity | 1 year
  Intensity of effort will be evaluated through the subjective perception of exertion scale. The scale goes from 1 to 10 values, and the closer to 10 the activity requires maximum effort, it seems almost impossible to continue.
Level of satisfaction | 1 year
  The level of satisfaction will be evaluated through the Physical Activity Enjoyment Scale. Scale from 1 to 7 values, the closer to 7 the more positive the physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina A Cabo, Principal Investigator — University of Évora
Locations (1):
- Carolina Alexandra Cabo, Evora, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bacha, J. M. R., Cordeiro, L. R., Alvisi, T. C., & Bonfim, T. R. (2016). Impacto do treinamento sensório-motor com plataforma vibratória no equilíbrio e na mobilidade funcional de um indivíduo idoso com sequela de acidente vascular encefálico: Relato de caso. Fisioterapia e Pesquisa, 23(1), 111-116. https://doi.org/10.1590/1809-2950/14362423012016
- [Background] Costa, J. N., Avelar, B. P., Gonçalves, C. D., & Pereira, M. M. (2012). Efeitos do circuito de equilíbrio sobre o equilíbrio funcional e a possibilidade de quedas em idosas. Motricidade, 8, 485-492.
- [Background] Gerhardy T, Gordt K, Jansen CP, Schwenk M. Towards Using the Instrumented Timed Up-and-Go Test for Screening of Sensory System Performance for Balance Control in Older Adults. Sensors (Basel). 2019 Feb 1;19(3):622. doi: 10.3390/s19030622. PMID 30717202
- [Background] Gléria, P. D. M. P., & Sandoval, R. A. (2011). Treinamento funcional como recurso fisioterapêutico para o aprimoramento da força muscular e equilíbrio de idosos. EFDeportes.com, Revista Digital, 161.
- [Background] Martins, M. M., Monteiro, C., Martinho, J., Guerra-Martín, M. D., Alves, I., & Vieira, M. (2016). Atividade física nos mais de 65 anos e a Promoção da Saúde. Actas de Gerontologia, 2(1).
- [Background] McGarrigle L, Boulton E, Todd C. Map the apps: a rapid review of digital approaches to support the engagement of older adults in strength and balance exercises. BMC Geriatr. 2020 Nov 18;20(1):483. doi: 10.1186/s12877-020-01880-6. PMID 33208117
- [Background] Pierratos, T., & Polatoglou, H. M. (2020). Utilizing the phyphox app for measuring kinematics variables with a smartphone. Physics Education, 55(2), 025019. https://doi.org/10.1088/1361-6552/ab6951
- [Background] Ready, E. A. (2019). Optimizing Gait Outcomes in Parkinson's Disease with Auditory Cues: The Effects of Synchronization, Groove, and Beat Perception Ability [The University of Western Ontario]. https://ir.lib.uwo.ca/etd
- [Background] Rezende, A. A. B., Silva, I. L. e, Beresford, H., & Batista, L. A. (2012). Avaliação dos efeitos de um programa sensório-motor no padrão da marcha de idosas. Fisioterapia em Movimento, 25(2), 317-324. https://doi.org/10.1590/S0103-51502012000200009
- [Background] Rikli, R. E., & Jones, C. J. (1999). Development and Validation of a Functional Fitness Test for Community-Residing Older Adults. Journal of Aging and Physical Activity, 7(2), 129-161. https://doi.org/10.1123/japa.7.2.129
- [Background] Rosa, B. P. de. S. (2012). Envelhecimento, Força Muscular e Atividade Física: Uma breve revisão bibliográfica. Revista Científica FacMais, 2(1), 140-152.
- [Background] Salehi, R., Ebrahimi-Takamjani, I., Esteki, A., Maroufi, N., & Parnianpour, M. (2010). Test-retest reliability and minimal detectable change for center of pressure measures of postural stability in elderly subjects. Medical Journal of the Islamic Republic of Iran, 23(4), 224-232.
- [Background] Sampaio, L. V. P., Castilho, L. B., & Carvalho, G. de A. (2017). Development of an application for mobile devices to evaluate the balance and risk of falls of the elderly. Revista Brasileira de Geriatria e Gerontologia, 20(6), 805-813. https://doi.org/10.1590/1981-22562017020.170017
- [Background] Serviço Nacional de Saúde. (2017). Tropeções, quedas e trambolhões. https://www.sns.gov.pt/noticias/2017/12/19/tropecoes-quedas-e-trambolhoes/
- [Background] Serviço Nacional de Saúde. (2018). Portal da Direção Nacional de Saúde. https://www.dgs.pt/programa-nacional-para-a-promocao-da-atividade-fisica/perguntas-e-respostas.aspx
- [Background] Suzuki, K., Niitsu, M., Kamo, T., Otake, S., & Nishida, Y. (2019). Effect of Exercise with Rhythmic Auditory Stimulation on Muscle Coordination and Gait Stability in Patients with Diabetic Peripheral Neuropathy: A Randomized Controlled Trial. Open Journal of Therapy and Rehabilitation, 07(03), 79-91. https://doi.org/10.4236/ojtr.2019.73005